CLINICAL TRIAL: NCT06850935
Title: Evaluation of the Skin Care Effects of Kristen Claire Supreme Rejuvenation Essence
Brief Title: Evaluation of Effects on Skin Quality of a Centella Asiatica Extracellular Vesicle-based Skin Care Formulation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hungkuang University (Other)
Responsible Party: Principal Investigator, Tsong-Min Chang, Vice President, Hungkuang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-064-A
Record Dates: First submitted 2025-02-26; First posted 2025-02-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Skin Quality; Skin Wrinkles; Melanin Hyperpigmentation; Skin Hydration; Skin Elasticity; Skin Redness
Keywords: Centella asiatica; Extracellular vesicles; Antioxidants; Cosmetics; Skin care; Anti-inflammatory; Skin whitening; UV damage; Photoaging; skin quality; gotu kola
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Centella asiatica extracellular vesicle formulation (Experimental): Water-based formulation containing purified Centella asiatica extracellular vesicle as main active ingredient.
  Interventions: Other: Centella asiatica extracellular vesicle formulation

INTERVENTIONS:
Other: Centella asiatica extracellular vesicle formulation — Water-based formulation containing purified Centella asiatica extracellular vesicle as main active ingredient. Applied twice daily at two drops per use to the face after face cleansing for 28 consecutive days.

SUMMARY:
The study evaluates the effects of a skin care formulation containing Centella asiatica extracellular vesicles as the main active ingredient on facial appearance and skin quality in healthy participants.

DETAILED DESCRIPTION:
Twenty healthy participants will be enrolled and will first undergo a 24-hour skin patch test on the forearm to assess potential irritation or allergic reactions to the test product. After screening, participants were asked to use the test product twice daily (morning and evening) after cleansing their face without using exfoliating products for 28 consecutive days. Each application involved 2 drops, evenly applied to the face using fingertips for absorption. Product usage was self-recorded, and the products were stored at room temperature.

The skin quality tests were conducted at the investigation site Hungkuang University onsite by the principal investigator. Each participant was to allocate 1 hour per test (including cleansing and waiting time). Skin quality tests were performed as a baseline test on day 0 (before using the test product), and subsequent tests at 7, 14, 21, and 28 days after test product use.

Measured parameters during assessment will include skin hydration, melanin content, skin elasticity, wrinkle percentage, redness area percentage, and pore percentage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of any gender from the age of 18 to 60 years (inclusive).
* Absence of chronic diseases, major illnesses, or allergies.

Exclusion Criteria:

* Currently using any medications or other skincare products

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Change in skin hydration | Assessment conducted every 7 days including Day 0 from Day 0 to Day 28 after treatment
  To measure skin hydration from Day 0 Day 28 of the study using C+K Multi Probe Adaptor MPA580 system with Corneometer CM825 Data probe, which evaluates the dielectric constant related to epidermal moisture at a depth of 60-100 µm. Data will be expressed as percentage of change in skin hydration relative to Day 0.
Change in skin melanin content | Assessment conducted every 7 days including Day 0 from Day 0 to Day 28 after treatment
  To measure skin melanin content from Day 0 Day 28 of the study using C+K Multi Probe Adaptor MPA580 system with Mexameter MX18 probe, which measures melanin and hemoglobin content using RGB light absorption at wavelengths 568 nm, 660 nm, and 880 nm. Data will be expressed as percentage of change in skin melanin content relative to Day 0.
Change in skin elasticity | Assessment conducted every 7 days including Day 0 from Day 0 to Day 28 after treatment
  To measure skin elasticity from Day 0 Day 28 of the study using C+K Multi Probe Adaptor MPA580 system with Cutometer Dual MPA580 probe by measuring skin stretching properties using suction-based method. Data will be expressed as percentage of change in skin elasticity relative to Day 0.
Change in skin wrinkle percentage | Assessment conducted every 7 days including Day 0 from Day 0 to Day 28 after treatment
  To measure skin elasticity from Day 0 Day 28 of the study using VISIA Skin Analysis System by using standard white light to detect shadow variations to determine the distribution and number of wrinkles. Fewer wrinkles yield higher percentages. Data will be expressed as percentage of change in skin wrinkle percentage relative to Day 0.
Change in skin redness percentage | Assessment conducted every 7 days including Day 0 from Day 0 to Day 28 after treatment
  To measure skin elasticity from Day 0 Day 28 of the study using VISIA Skin Analysis System by using RBX polarized light to identify vascular or inflammatory issues. Smaller red zones result in higher percentages. Data will be expressed as percentage of change in skin redness percentage relative to Day 0.
Change in skin pore percentage | Assessment conducted every 7 days including Day 0 from Day 0 to Day 28 after treatment
  To measure skin elasticity from Day 0 Day 28 of the study using VISIA Skin Analysis System by using white light to analyze shadowed pore depressions and darker areas relative to surrounding skin. Fewer pores yield higher percentages. Data will be expressed as percentage of change in skin pore percentage relative to Day 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Hungkuang University, Taichung, Taiwan